CLINICAL TRIAL: NCT01826019
Title: Heart Outcomes Prevention and Evaluation 4 (HOPE-4)
Brief Title: Heart Outcomes Prevention and Evaluation 4
Acronym: HOPE-4
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Population Health Research Institute (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Grand Challenges Canada (Other); Global Alliance for Chronic Diseases (GACD) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HOPE-4
Record Dates: First submitted 2013-03-31; First posted 2013-04-08 (Estimated); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Hypertension; Cardiovascular Disease
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Intensive CV risk detection, counselling and follow-up program by NPHW; recommended CV medications will include combinations of anti-hypertensive medications (both low and high doses) and a lipid lowering agent (e.g. statin) in accordance with treatment algorithm [precise formulations used may differ in each country]; use of treatment supporters to reinforce adherence.
  Interventions: Other: Intervention
- Control - Usual Care (Other): Participants in control communities will be referred to usual care.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Intervention — In intervention communities, management plans will be developed by the NPHW for all enrolled participants. The NPHWs will educate participants about CVD, HT treatment, lifestyle modifications and initiate therapy according to the modified WHO CVD risk-management algorithm, including referral of high-risk patients to physicians and safety monitoring where appropriate. Participants in intervention communities will have support from family or friends (treatment supporters) and will receive educational materials and treatment reminders using text-messaging, email, and printed materials, as appropriate for the participant and the community setting. Evidence-based CV medications will be made available to the NPHWs and supervising physicians for participant treatment.
  Arms: Intervention
Other: Usual Care — At initial screening, eligible participants will be provided with a brief information booklet/leaflet (customized to the community or region) regarding lifestyle modification and be advised to see their usual physician for care that is considered appropriate. No structured interventions will be employed.
  Arms: Control - Usual Care

SUMMARY:
The overall objective of the HOPE-4 Phases (HT and CVD) is to develop, implement and evaluate an evidence-based, contextually appropriate programme for cardiovascular disease (CVD) risk assessment, treatment and control involving: (1) simplified algorithms implemented by non-physician health workers (NPHW) and supported by e-health technologies (tablets programmed with decision and counselling support software); (2) initiation of evidence-based cardiovascular (CV) medications and (3) treatment supporters to optimize long-term medication and lifestyle adherence.

DETAILED DESCRIPTION:
Study design: open-label, parallel cluster randomized controlled trial design.

HT Phase: Up to 30 urban and rural communities in Canada, Colombia and Malaysia will be randomized to participate in an intensive CV risk detection and control programme by NPHW or to care as usual for 12 months. NOTE: Canada will serve as a pilot study, which will be used to evaluate feasibility, time, cost and program improvements.

CVD Phase: If funded, this phase will be a continuation and expansion of HT Phase to include up to 190 urban and rural communities in countries within Asia, South America, Sub-Saharan Africa, and Canada that will be allocated to participate in an intensive CV risk detection and control programme supported by NPHWs or to care as usual for up to 6 years. NOTE: CVD Phase - currently not initiated.

Communities will be randomized 1:1 with a central randomization system to either a) intervention or b) control, after screening in the community is complete.

ELIGIBILITY:
Inclusion Criteria:

Individuals (≥ 50 years) with at least ONE of the following criteria:

1. SBP ≥160 mmHg in one visit
2. SBP 140-159 mmHg in one visit AND participant-reported medical diagnosis of hypertension
3. SBP 140-159 mmHg in one visit AND participant taking anti-HT medication
4. SBP ≥130 mmHg in one visit AND participant-reported medical diagnosis of diabetes
5. SBP ≥130 mmHg in one visit AND participant taking medication for diabetes
6. Participants that do not meet criteria 1-5 AND SBP 140-159 mmHg in one visit AND SBP ≥140 mmHg in a second visit ≥24 hours apart

Exclusion Criteria:

1. Refusal to Consent
2. Actively involved in any study or heart health program that would compromise the protocol of HOPE-4
3. Severe co-morbid condition with life expectancy < 1 year
4. Other serious condition(s) or logistic factors likely to interfere with study participation or with the ability to complete the trial, as appropriate to country or region.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1438 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
The mean difference in change in Framingham Risk Score (FRS) between the intervention and control communities from baseline to 1 year. | Baseline to 1 year (HT phase)
Difference in major CV events [CV death, CV hospitalizations (e.g. MI, Stroke, AF, unstable or new onset angina, CHF, arterial revascularization), and end-stage renal disease] at 6 years. | Undetermined - currently not initiated and is dependent on funding (CVD Phase).

SECONDARY OUTCOMES:
Change in systolic BP (SBP) between the intervention and control communities at 6 and 12 months | Baseline to 6 months and 12 months (HT Phase)
Proportion of participants with well-controlled blood pressure at 6 and 12 months (SBP < 140 mmHg in non-diabetics and SBP < 130 mmHg in diabetics | Baseline to 6 months and 12 months (HT Phase)
Change in HDL, LDL, total cholesterol, triglycerides, and glucose levels at 12 months | Baseline to 1 year (HT Phase)
Change in smoking status at 6 and 12 months | Baseline to 6 months and 12 months (HT Phase)
Change in IHRS at 6 and 12 months and ChRS at 12 months | Baseline to 6 months and 12 months (HT Phase)
Number of participants receiving prescriptions for (or taking) anti-hypertensive medications (as an indication of physician adherence to treatment guidelines) at 6 and 12 months | Baseline to 6 months and 12 months (HT Phase)
Medication adherence measures at 6 and 12 months | Baseline to 6 months and 12 months (HT Phase)
Clinical events (e.g. death, CVD development, hospitalizations) at 6 and 12 months | Baseline to 6 months and 12 months (HT Phase)
Country-specific process outcomes at 6 and 12 months | Baseline to 6 months and 12 months (HT Phase)
Change in individual components of the primary outcomes in the HT Phase | Undetermined - currently not initiated and is dependent on funding (CVD Phase)
Secondary outcomes from the HT Phase | Undetermined - currently not initiated and is dependent on funding (CVD Phase)

OTHER OUTCOMES:
A descriptive analysis of the processes involved in the intervention | Baseline to 1 year
Qualitative feedback from participants, NPHWs, and supervising physicians | Baseline to 1 year
Health economic and quality of life evaluations (as available and appropriate). | Baseline to 1 year
  We will collect data that will allow us to determine (i) the costs of the suggested programs (i.e. intervention package) and the costs of what is being provided currently for CVD assessment and management in the communities studied (i.e. control).

CONTACTS AND LOCATIONS:
Overall Officials: Jon-David Schwalm, MD, MSc, Principal Investigator — McMaster University and Hamilton Health Sciences Corp.; Salim Yusuf, MD, DPhil, Principal Investigator — McMaster University and Hamilton Health Sciences Corp.
Locations (4):
- Canada (2):
  - Simon Fraser University, Burnaby, British Columbia
  - Population Health Research Institute, Hamilton, Ontario
- FOSCAL, Floridablanca, Santander Department, Colombia
- UniversitiTeknologi MARA (UiTM), Sungai Buloh, Selangor, Malaysia

REFERENCES:
- [Derived] Drakos A, McCready T, Lopez-Jaramillo P, Islam S, McKee M, Yusuf S, Schwalm JD. Relationship Between Social Support and Clinical Outcomes: An Evaluation of Participant-Nominated Treatment Supporters in the HOPE 4 Intervention. Circ Cardiovasc Qual Outcomes. 2024 Apr;17(4):e009342. doi: 10.1161/CIRCOUTCOMES.122.009342. Epub 2024 Mar 5. PMID 38440889
- [Derived] Schwalm JD, McCready T, Lopez-Jaramillo P, Yusoff K, Attaran A, Lamelas P, Camacho PA, Majid F, Bangdiwala SI, Thabane L, Islam S, McKee M, Yusuf S. A community-based comprehensive intervention to reduce cardiovascular risk in hypertension (HOPE 4): a cluster-randomised controlled trial. Lancet. 2019 Oct 5;394(10205):1231-1242. doi: 10.1016/S0140-6736(19)31949-X. Epub 2019 Sep 2. PMID 31488369
- [Derived] Schwalm JR, McCready T, Lamelas P, Musa H, Lopez-Jaramillo P, Yusoff K, McKee M, Camacho PA, Lopez-Lopez J, Majid F, Thabane L, Islam S, Yusuf S. Rationale and design of a cluster randomized trial of a multifaceted intervention in people with hypertension: The Heart Outcomes Prevention and Evaluation 4 (HOPE-4) Study. Am Heart J. 2018 Sep;203:57-66. doi: 10.1016/j.ahj.2018.06.004. Epub 2018 Jun 22. PMID 30015069
- See also: Population Health Research Institute — http://www.phri.ca